CLINICAL TRIAL: NCT06602063
Title: Surgery With ICBs in BRCAwt, CD8+ TILs, 1st Relapsed Ovarian Cancer: A Pilot Study
Brief Title: Surgery for Relapsed Ovarian Cancer in Precision
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Gynecologic Oncology Group (Other Government)
Collaborators: Shanghai Zhongshan Hospital (Other); Tongji Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOC-P
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: Ovarian cancer; Immune checkpoint inhibitor; Secondary cytoreduction; Biomarker-driven
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Surgical Procedures, Operative; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- criteria-fulfilled arm (Experimental): Patients who meet the inclusion and exclusion criteria will receive secondary cytoreductive surgery followed by 6 cycles of post-operative chemotherapy with Iparomlimab/tuvonralimab maintenance therapy.
  Interventions: Procedure: surgery/chemotherapy; Drug: Iparomlimab/Tuvonralimab
- compassionate use arm (Experimental): Patients who are enrolled under expanded eligibility criteria will receive secondary cytoreductive surgery followed by 6 cycles of post-operative chemotherapy with Iparomlimab/tuvonralimab maintenance therapy.
  Interventions: Procedure: surgery/chemotherapy; Drug: Iparomlimab/Tuvonralimab
- real world arm (No Intervention): Patients who meet the inclusion and exclusion criteria but refuse to participate in the CF and CU arms will receive the physician's therapy of choice.

INTERVENTIONS:
Procedure: surgery/chemotherapy — secondary cytoreductive surgery followed by 6 cycles of post-operative chemotherapy
  Arms: compassionate use arm; criteria-fulfilled arm
Drug: Iparomlimab/Tuvonralimab — Iparomlimab/tuvonralimab will be administered at a dose of 5 mg per kilogram IV every 21 days. Treatment will continue until disease progression confirmed by RECIST criteria v1.1, intolerable toxicity or withdrawal of consent.
  Arms: compassionate use arm; criteria-fulfilled arm

SUMMARY:
This multicenter, biomarker-driven, patient-centric study aimed to evaluate the efficacy of secondary cytoreduction followed by platinum-based chemotherapy in combination with anti-PD1/CTLA-4 bispecifics therapy in patients with platinum-sensitive relapsed ovarian cancer (PSROC).

DETAILED DESCRIPTION:
The immune phenotype of patients with relapsed ovarian cancer may correlate with their response to immunotherapy. This multicenter, biomarker-driven, patient-centric study aimed to evaluate the efficacy of secondary cytoreduction followed by platinum-based chemotherapy in combination with anti-PD1/CTLA-4 bispecifics therapy in patients with platinum-sensitive relapsed ovarian cancer (PSROC). PD-L1 expression and CD8+ tumor-infiltrating T cell count (CD8+ TILs count) were evaluated as biomarkers using archived or fresh tumor tissue samples in patients with BRCA1/2 wild type.

This study would be proceeded in two phases. The phase 1b single-arm study aimed to evaluate the efficacy of Iparomlimab/tuvonralimab in the treatment of BRCA wild type, PD-L1-positive, CD8+ TILs-positive, patients with PSROC. The patent-centric phase II study with three arms aimed to evaluate the efficacy of secondary cytoreduction followed by platinum-based chemotherapy in combination with Iparomlimab/tuvonralimab in these patients. In arm 1 and 2, patients received secondary cytoreduction followed by platinum-based chemotherapy in combination with Iparomlimab/tuvonralimab. In arm 3, patients received physician's therapy of choice.

ELIGIBILITY:
Inclusion Criteria:

* Arm 1 (criteria-fulfilled, CF)

  1. Age at recurrence ≥ 18 years, <80 years.
  2. Patients with platinum-sensitive, first relapsed epithelial ovarian, primary peritoneal, or fallopian tube cancer (EOC, PPC, FTC), which is defined as those with treatment -free interval of 6 months or more.
  3. If the patient had previous PARPi maintenance therapy, disease progression should occurring at lease 3 months after the prior PARPi withdrawal.
  4. BRCA1/2 wild type (both germline and somatic)
  5. Homologous Recombination Deficiency (HRD) is available
  6. Patients must provide archived or fresh tumor tissue samples for biomarker detection.
  7. PD-L1 positive (if either at least 1% of assessed tumour cells expressed membranous PD-L1, at least 5% of immune cells within the tumour area expressed PD-L1, or both) and number of intraepithelial CD8+ tumor-infiltrating lymphocytes (TILs) per high-powered field ≥ 6.
  8. Assessed by the experienced surgeons, complete resection of all recurrent disease is possible (predicted by iMODEL score or by PET/CT).
  9. ECOG performance status of 0 to 2
  10. Adequate bone marrow, liver, and renal function to receive combined immunotherapy
  11. Written informed consent
* Arm 2 (compassionate use, CU), Similar to cohort 1, except for:

  1. If the patient had previous PARPi maintenance therapy, disease progression should occurring within 3 months after the prior PARPi withdrawal or during the PARPi maintenance therapy.
  2. PD-L1 positive or number of intraepithelial CD8+ TILs per high-powered field ≥ 6.
* Arm 3 (real word) Patients who meet the inclusion criteria but refuse to participate in the phase II CF and CU cohorts.

Exclusion Criteria:

1. Patients with borderline, low-grade tumors, clear cell carcinoma, as well as non-epithelial tumors.
2. Patients with platinum-resistant or refractory diseases.
3. Lack of tumor samples (archived and/or recently obtained) for biomarker detection.
4. Previous administration of immunotherapy
5. Patients have been vaccinated with the live vaccine or received anti-tumor treatment within 4 weeks before the first administration.
6. Synchronous or metachronous (within 5 years) malignancy, symptomatic or uncontrolled visceral metastases that require simultaneous treatment, other than carcinoma in situ or breast cancer (without any signs of relapse or activity).
7. Patients with parenchymal metastases and life-threatening complications in short term.
8. Any other concurrent medical conditions contraindicating surgery, chemotherapy, or immunotherapy that could compromise the adherence to the protocol.
9. Patients are known to be allergic to the active ingredients or excipients of Sintilimab.
10. HRD status is not available.
11. Any medication induced considerable risk of surgery, e.g. estimated bleeding due to oral anticoagulating agents or bevacizumab.
12. Patients for interval-debulking, or for second-look surgery, or palliative surgery planned.
13. Impossible to assess the resectability of recurrent disease or evaluate the score. Radiological signs suggesting complete resection is impossible.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — participant eligibility is based on self-representation of gender identity
Enrollment: 33 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival in CF arm | Up to 3 years
  The time from entry into the study to the diagnosis of the first progression or recurrence or death in CF arm, whichever occurs first
3-years Overall Survival Rate in CF arm | Up to 3 years
  The proportion of patients without death at 3 years after entry into the study in CF arm

SECONDARY OUTCOMES:
Overall survival in CF arm | Up to 3 years
  The time from entry into the study to the date of death from any cause or last follow-up in CF arm
TFST in CF arm | Up to 3 years
  Time from entry into the study until the starting date of the first subsequent anticancer therapy or death, whichever occurred first, whichever occurred first, in CF arm
TSST in CF arm | Up to 3 years
  Time from entry into the study until the starting date of the second subsequent anticancer therapy or death, whichever occurred first, in CF arm
Post-operative complications in CF and CU arms | Up to 1 months
  The surgical complications will be evaluated at 30-day after secondary cytoreductive surgery in CF and CU arms
Quality of life assessments in CF arm using EORTC QLQ-C30 | Up to 3 years
  Changes in EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30) scores in CF arm (baseline; 6 months, 12 months, 24 months and 36 months after entry into the study; score range 0-126; higher score = worse outcome)
Quality of life assessments in CF arm using FACT-O | Up to 3 years
  Changes in FACT-O (Functional Assessment of Cancer Therapy-Ovarian cancer) scores in CF arm (baseline; 6 months, 12 months, 24 months and 36 months after entry into the study; score range 0-156; higher score = worse outcome)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhongshan Hospital Fudan University, Shanghai
  - Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: No